CLINICAL TRIAL: NCT01762423
Title: PEMF Effects on Pain After Abdominal Body Contouring
Acronym: PEMF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding issues.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO12070504
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Abdominal Body Contouring Surgery; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Device (Experimental): Device Placement:
  Upon completion of the subjects' standard of care body contouring surgery, the device will be placed directly on the operative dressings within an unobtrusive binder with Velcro strips and will be activated before the subject leaves the OR. Subjects will then be educated on the functionality and interpretation of the user interface of the device. They will be educated on the application, removal, and return of the device.
  Active Devices The device will be activated at the time of placement. The active devices are programmed to automatically deliver treatment. Each treatment duration is 15 minutes. The active device delivers treatment every 2 hours. A light will flash on the device when the PEMF begins and will continue to flash every second until the end of the treatment. Between treatments the device will be in "sleep mode" and the light will flash every 5 seconds.
  Interventions: Device: Active Device (IVIVI SofPulse)
- Sham Device (Sham Comparator): Device Placement:
  Upon completion of the subjects' standard of care body contouring surgery, the device will be placed directly on the operative dressings within an unobtrusive binder with velcro strips and will be activated before the subject leaves the OR. Subjects will then be educated on the functionality and interpretation of the user interface of the device. They will be educated on the application, removal, and return of the device.
  Sham Devices The sham devices mirror the active device with the exception of the delivery of the PEMF. The sham device will be "activated" at the time of placement. A light will flash on the device when the SHAM PEMF begins and will continue to flash every second until the end each treatment interval. While in "sleep mode" the device will not deliver treatment and the light will flash every 5 seconds.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Active Device (IVIVI SofPulse)
  Other Names: IVIVI SofPulse
  Arms: Active Device
Device: Sham Device
  Arms: Sham Device

SUMMARY:
Body contouring surgery has a higher potential for postoperative pain and wound healing complications. The purpose of this study is to determine if pulsed electromagnetic field (PEMF) devices can reduce the pain and complications associated with this type of surgery.

Pulsed electromagnetic field (PEMF) devices have been shown to be effective treatments to decrease healing time in nonunion fractures and pressure ulcers, and to reduce pain in whiplash injuries, persistent neck pain, and chronic lower back pain. These devices have been FDA approved for treatment of pain and edema (510(k) number: K070541). More recently, PEMF devices have been shown to decrease postoperative pain and narcotic use in breast augmentation patients. This study seeks to determine if PEMF will also cause similar effects in the more complex procedures performed on body contouring patients. The specific aims of this study are:

1. Evaluate if adjunct PEMF therapy will accelerate the rate of postoperative pain reduction in abdominal body contouring patients.
2. Evaluate if adjunct PEMF therapy will decrease the postoperative use of narcotic pain relievers in abdominal body contouring patients.

PEMF devices have been shown to be effective in reduction of pain and pain medication use in breast augmentation patients. No literature has shown if PEMF is an effective adjunct to decrease pain or pain medication use in the abdominal body contouring patient. A decrease in pain would result in a better experience for patients and a reduction in pain medication may decrease complications associated with these medications. The PEMF therapy device being used in this study is a non-significant risk device because it is noninvasive and does not present a potential for serious risk to the health, safety, or welfare of a subject.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older and able to provide informed consent
* Eligible for and have agreed to be scheduled for elective abdominal body contouring surgery
* Willing and able to comply with all study procedures.

Exclusion Criteria:

* Inability to provide informed consent
* Patients having multiple procedures concurrently except liposuction.
* Current use of oral steroids as determined through patient history and medical record review
* Current narcotic use as determined through patient history or medical record review
* Current nerve or pain disorder.
* Recent (1 month) coronary stent or implanted medical device (e.g. pacemaker).
* Pregnancy (demonstrated by a positive result of a urine pregnancy test)
* Based upon surgeon judgement and the results of screening procedures, patient is not a suitable candidate for surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Reduction | Immediately postoperatively through 6 days postoperative
  Evaluate if adjunct PEMF therapy will accelerate the rate of postoperative pain reduction in abdominal body contouring patients.

SECONDARY OUTCOMES:
Postoperative Narcotic Use | Immediately postoperative through 6 day postoperative
  Evaluate if adjunct PEMF therapy will decrease the postoperative use of narcotic pain relievers in abdominal body contouring patients.

CONTACTS AND LOCATIONS:
Overall Officials: J. Peter Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Center for Innovation in Restorative Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Akai M, Hayashi K. Effect of electrical stimulation on musculoskeletal systems; a meta-analysis of controlled clinical trials. Bioelectromagnetics. 2002 Feb;23(2):132-43. doi: 10.1002/bem.106. PMID 11835260
- [Background] Akai M, Kawashima N, Kimura T, Hayashi K. Electrical stimulation as an adjunct to spinal fusion: a meta-analysis of controlled clinical trials. Bioelectromagnetics. 2002 Oct;23(7):496-504. doi: 10.1002/bem.10041. PMID 12224053
- [Background] Griffin XL, Warner F, Costa M. The role of electromagnetic stimulation in the management of established non-union of long bone fractures: what is the evidence? Injury. 2008 Apr;39(4):419-29. doi: 10.1016/j.injury.2007.12.014. Epub 2008 Mar 5. PMID 18321512
- [Background] Heden P, Pilla AA. Effects of pulsed electromagnetic fields on postoperative pain: a double-blind randomized pilot study in breast augmentation patients. Aesthetic Plast Surg. 2008 Jul;32(4):660-6. doi: 10.1007/s00266-008-9169-z. Epub 2008 May 28. PMID 18506512
- [Background] Greco JA 3rd, Castaldo ET, Nanney LB, Wendel JJ, Summitt JB, Kelly KJ, Braun SA, Hagan KF, Shack RB. The effect of weight loss surgery and body mass index on wound complications after abdominal contouring operations. Ann Plast Surg. 2008 Sep;61(3):235-42. doi: 10.1097/SAP.0b013e318166d351. PMID 18724119
- [Background] Coon D, Gusenoff JA, Kannan N, El Khoudary SR, Naghshineh N, Rubin JP. Body mass and surgical complications in the postbariatric reconstructive patient: analysis of 511 cases. Ann Surg. 2009 Mar;249(3):397-401. doi: 10.1097/SLA.0b013e318196d0c6. PMID 19247025
- [Background] Nagai M, Ota M. Pulsating electromagnetic field stimulates mRNA expression of bone morphogenetic protein-2 and -4. J Dent Res. 1994 Oct;73(10):1601-5. doi: 10.1177/00220345940730100401. PMID 7929974
- [Background] Liboff AR, Williams T Jr, Strong DM, Wistar R Jr. Time-varying magnetic fields: effect on DNA synthesis. Science. 1984 Feb 24;223(4638):818-20. doi: 10.1126/science.6695183.
- [Background] Ozawa H, Abe E, Shibasaki Y, Fukuhara T, Suda T. Electric fields stimulate DNA synthesis of mouse osteoblast-like cells (MC3T3-E1) by a mechanism involving calcium ions. J Cell Physiol. 1989 Mar;138(3):477-83. doi: 10.1002/jcp.1041380306. PMID 2538484
- [Background] Miura M, Takayama K, Okada J. Increase in nitric oxide and cyclic GMP of rat cerebellum by radio frequency burst-type electromagnetic field radiation. J Physiol. 1993 Feb;461:513-24. doi: 10.1113/jphysiol.1993.sp019526. PMID 7688808
- [Background] Diniz P, Soejima K, Ito G. Nitric oxide mediates the effects of pulsed electromagnetic field stimulation on the osteoblast proliferation and differentiation. Nitric Oxide. 2002 Aug;7(1):18-23. doi: 10.1016/s1089-8603(02)00004-6. PMID 12175815
- [Background] Witte MB, Thornton FJ, Efron DT, Barbul A. Enhancement of fibroblast collagen synthesis by nitric oxide. Nitric Oxide. 2000 Dec;4(6):572-82. doi: 10.1006/niox.2000.0307. PMID 11139365
- [Background] Liboff AR, Cherng S, Jenrow KA, Bull A. Calmodulin-dependent cyclic nucleotide phosphodiesterase activity is altered by 20 microT magnetostatic fields. Bioelectromagnetics. 2003 Jan;24(1):32-8. doi: 10.1002/bem.10063. PMID 12483663
- [Background] Korhonen R, Lahti A, Kankaanranta H, Moilanen E. Nitric oxide production and signaling in inflammation. Curr Drug Targets Inflamm Allergy. 2005 Aug;4(4):471-9. doi: 10.2174/1568010054526359. PMID 16101524
- [Background] Reale M, De Lutiis MA, Patruno A, Speranza L, Felaco M, Grilli A, Macri MA, Comani S, Conti P, Di Luzio S. Modulation of MCP-1 and iNOS by 50-Hz sinusoidal electromagnetic field. Nitric Oxide. 2006 Aug;15(1):50-7. doi: 10.1016/j.niox.2005.11.010. Epub 2006 Feb 7. PMID 16455275
- [Background] Jeong JH, Kum C, Choi HJ, Park ES, Sohn UD. Extremely low frequency magnetic field induces hyperalgesia in mice modulated by nitric oxide synthesis. Life Sci. 2006 Feb 23;78(13):1407-12. doi: 10.1016/j.lfs.2005.07.006. Epub 2006 Feb 7. PMID 16457856
- [Background] Fitzsimmons RJ, Gordon SL, Kronberg J, Ganey T, Pilla AA. A pulsing electric field (PEF) increases human chondrocyte proliferation through a transduction pathway involving nitric oxide signaling. J Orthop Res. 2008 Jun;26(6):854-9. doi: 10.1002/jor.20590. PMID 18240331
- [Background] Pilla AA, Nasser PR, Kaufman JJ. Gap junction impedance, tissue dielectrics and thermal noise limits for electromagnetic field bioeffects. Bioelectrochem Bioenerg (1994) 35:63-69
- [Background] Strauch B, Patel MK, Rosen DJ, Mahadevia S, Brindzei N, Pilla AA. Pulsed magnetic field therapy increases tensile strength in a rat Achilles' tendon repair model. J Hand Surg Am. 2006 Sep;31(7):1131-5. doi: 10.1016/j.jhsa.2006.03.024. PMID 16945715
- [Background] Strauch B, Patel MK, Navarro JA, Berdichevsky M, Yu HL, Pilla AA. Pulsed magnetic fields accelerate cutaneous wound healing in rats. Plast Reconstr Surg. 2007 Aug;120(2):425-430. doi: 10.1097/01.prs.0000267700.15452.d0. PMID 17632344
- [Background] Roland D, Ferder M, Kothuru R, Faierman T, Strauch B. Effects of pulsed magnetic energy on a microsurgically transferred vessel. Plast Reconstr Surg. 2000 Apr;105(4):1371-4. doi: 10.1097/00006534-200004040-00016. PMID 10744227
- [Background] Gilbert TL, Griffin N, Moffett J, Ritz MC, George FR. The Provant Wound Closure System induces activation of p44/42 MAP kinase in normal cultured human fibroblasts. Ann N Y Acad Sci. 2002 Jun;961:168-71. doi: 10.1111/j.1749-6632.2002.tb03076.x. No abstract available. PMID 12081892
- [Background] Callaghan MJ, Chang EI, Seiser N, Aarabi S, Ghali S, Kinnucan ER, Simon BJ, Gurtner GC. Pulsed electromagnetic fields accelerate normal and diabetic wound healing by increasing endogenous FGF-2 release. Plast Reconstr Surg. 2008 Jan;121(1):130-141. doi: 10.1097/01.prs.0000293761.27219.84. PMID 18176216
- [Background] Gardner SE, Frantz RA, Schmidt FL. Effect of electrical stimulation on chronic wound healing: a meta-analysis. Wound Repair Regen. 1999 Nov-Dec;7(6):495-503. doi: 10.1046/j.1524-475x.1999.00495.x. PMID 10633009
- [Background] Stiller MJ, Pak GH, Shupack JL, Thaler S, Kenny C, Jondreau L. A portable pulsed electromagnetic field (PEMF) device to enhance healing of recalcitrant venous ulcers: a double-blind, placebo-controlled clinical trial. Br J Dermatol. 1992 Aug;127(2):147-54. doi: 10.1111/j.1365-2133.1992.tb08047.x. PMID 1390143
- [Background] Tepper OM, Callaghan MJ, Chang EI, Galiano RD, Bhatt KA, Baharestani S, Gan J, Simon B, Hopper RA, Levine JP, Gurtner GC. Electromagnetic fields increase in vitro and in vivo angiogenesis through endothelial release of FGF-2. FASEB J. 2004 Aug;18(11):1231-3. doi: 10.1096/fj.03-0847fje. Epub 2004 Jun 18. PMID 15208265